CLINICAL TRIAL: NCT02757677
Title: A Cross-sectional, Prospective, Observational Study to Evaluate Blood Flow Characteristics in Glaucoma Patients Using Optical Coherence Tomography Based Angiography (OCT-A).
Brief Title: Evaluation of Blood Flow Characteristics in Glaucoma Using Optical Coherence Tomography Angiography (OCT-A).
Status: Terminated | Type: Observational
Why Stopped: Difficulties with recruitment
Sponsor: Swiss Vision Network (Other)
Responsible Party: Principal Investigator, Dr. Kaweh Mansouri, dr. Kaweh Mansouri, Swiss Vision Network
Other Study IDs: GR-02
Record Dates: First submitted 2016-04-13; First posted 2016-05-02 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Longitudinal arm: Evaluate optic nerve head blood flow using the new OCT-A software in surgically and medically treated glaucoma patients and in different types of glaucoma
  Interventions: Device: Optical Coherence Tomography based Angiography
- 24-h Intraocular pressure (IOP) arm: Evaluate the correlation between circadian IOP changes and optic nerve head blood flow using the new OCT-A software
  Interventions: Device: Optical Coherence Tomography based Angiography
- Surgery arm: Evaluate blood flow using the new OCT-A software in surgically treated glaucoma patients
  Interventions: Device: Optical Coherence Tomography based Angiography

INTERVENTIONS:
Device: Optical Coherence Tomography based Angiography — A contrast-free, noninvasive technology to identify blood vessels in the eye

SUMMARY:
The investigators aim to evaluate the efficacy of the new Optical Coherence Tomography based Angiography (OCT-A) softwares in the diagnosis and management of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open angle glaucoma (OAG) including pseudo-exfoliative and pigmentary glaucoma.
* Documented glaucomatous visual field damage (in the previous 12 months with mean defect (MD) > 2.0 dB)
* Structural and/or functional glaucomatous damage
* Have given written informed consent, prior to any investigational procedures

Exclusion Criteria:

* Patients with allergy to corneal anesthetic
* Patients not able to understand the character and individual consequences of the investigation
* Participation in other clinical research within the last 4 weeks
* Other diseases that may cause visual field loss or optic disc abnormalities
* Refractive error of > +3.00D or < -7.00D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be enrolled from glaucoma clinics of the Montchoisi glaucoma center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Macular and optic nerve head bloodflow, as measured by OCT-A macular and optic nerve head vessel density (%) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kaweh Mansouri, MD, Principal Investigator — Glaucoma center, Montchoisi clinic, Swiss vision network
Locations (1):
- Glaucoma center, Montchoisi clinic, Lausanne, Switzerland